CLINICAL TRIAL: NCT00880737
Title: Prognostic Value of Computed Tomography (CT) Scan in Hemodynamically Stable Patients With Acute Symptomatic Pulmonary Embolism
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Carlos III Health Institute (Other Government)
Other Study IDs: FIS 2008
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stable PE patients: Hemodynamically stable patients with acute symptomatic pulmonary embolism

SUMMARY:
The objectives of the PROTECT study are:

* To assess the role of CT pulmonary angiography in the risk stratification of hemodynamically stable patients with acute symptomatic pulmonary embolism (PE).
* To assess the role of transthoracic echocardiography in the risk stratification of hemodynamically stable patients with acute symptomatic PE.
* To assess the role of 2 biomarkers (troponin and brain natriuretic peptide) in the risk stratification of hemodynamically stable patients with acute symptomatic PE.
* To assess the role of the Pulmonary Embolism Severity Index (PESI) in the risk stratification of hemodynamically stable patients with acute symptomatic PE.
* To assess the combined role of CT pulmonary angiography, transthoracic echocardiography, PESI, troponin I and brain natriuretic peptide in the risk stratification of hemodynamically stable patients with acute symptomatic PE.

ELIGIBILITY:
Inclusion Criteria:

* Acute symptomatic Pulmonary Embolism (PE) confirmed by:

  * CT pulmonary angiography positive for PE
  * Ventilation/ perfusion lung scan with high likelihood of PE (according to PIOPED criteria)
  * V/Q ventilation/ perfusion lung scan inconclusive for PE or negative CT pulmonary angiography in a patient with thoracic symptoms and a lower limb ultrasound showing a positive diagnosis for deep vein thrombosis.

Exclusion Criteria:

* Contraindication for CT pulmonary angiography (allergy to iodine contrasts or creatinin clearance < 30 ml/min).
* Informed consent not obtained.
* Pregnancy.
* Life expectancy of less than 3 months.
* Hemodynamic unstability defined as SBP < 90 mm Hg, need for cardiopulmonary reanimation, need for vasoactive drugs or orotracheal intubation.
* Thrombectomy, insertion of filter in the cava vein, or need for fibrinolytic treatment for PE episode.
* Participation in another clinical trial for treatment of PE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodynamically stable outpatients with suspicion of pulmonary embolism, confirmed by objective testing
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome considered will be death by any cause in the month following diagnosis. | 30 days after PE diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ramón y Cajal Hospital, Madrid, Spain

REFERENCES:
- [Derived] Lankeit M, Jimenez D, Kostrubiec M, Dellas C, Kuhnert K, Hasenfuss G, Pruszczyk P, Konstantinides S. Validation of N-terminal pro-brain natriuretic peptide cut-off values for risk stratification of pulmonary embolism. Eur Respir J. 2014 Jun;43(6):1669-77. doi: 10.1183/09031936.00211613. Epub 2014 Mar 13. PMID 24627529